CLINICAL TRIAL: NCT04926233
Title: Characteristics and Treatment Patterns of Patients With Chronic Obstructive Pulmonary Disease (COPD), Initiating Tio+Olo or Other Maintenance Therapies in the US and the UK: A Retrospective Claims Database Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0091
Record Dates: First submitted 2021-06-13; First posted 2021-06-15 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- COPD patients from US IBM Marketscan database
  Interventions: Drug: Tiotropium bromide + Olodaterol; Device: Sp(t)iolto® Respimat®
- COPD patients from UK CPRD GOLD database
  Interventions: Drug: Tiotropium bromide + Olodaterol; Device: Sp(t)iolto® Respimat®

INTERVENTIONS:
Drug: Tiotropium bromide + Olodaterol — Tiotropium bromide + Olodaterol
  Other Names: Sp(t)iolto® Respimat®
Device: Sp(t)iolto® Respimat® — Sp(t)iolto® Respimat®

SUMMARY:
The primary objectives of the study are to use US and UK data to describe the characteristics of Chronic Obstructive Pulmonary Disease (COPD) patients according to various demographic, lifestyle, clinical, and medication use.

ELIGIBILITY:
Inclusion criteria:

* parent cohort

  -- COPD diagnosis
* child cohort

  -- any initiation of first maintenance therapy after July 1, 2015
* grandchild cohort -- any initiation of second maintenance therapy after August 2, 2015

Exclusion criteria:

- parent cohort

* age <40 on index date
* any COPD diagnosis in baseline
* any use of long-acting muscarinic antagonists (LAMA), long-acting beta-agonists (LABA), or inhaled corticosteroid (ICS) in baseline
* <365 days of continuous medical and pharmacy coverage

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for the analysis will consist of all patients with at least one medical claim with a diagnosis code of COPD identified.
Sampling Method: Non-Probability Sample
Enrollment: 1371146 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AETION inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This retrospective cohort study used previously collected administrative healthcare data (United States data from IBM MarketScan and United Kingdom data from CPRD GOLD, a primary care database) to describe the patients characteristics and treatment patterns in patients with chronic obstructive pulmonary disease (COPD), initiating tiotropium + olodaterol or other maintenance therapies.
Pre-assignment Details: Patients with chronic obstructive pulmonary disease (COPD) who met all inclusion criteria and none of the exclusion criteria initiating tiotropium + olodaterol or other maintenance therapies from either IBM MarketScan (United States) or CPRD GOLD (United Kingdom) databases were included.
Groups:
- US IBM Marketscan - Overall: All chronic obstructive pulmonary disease (COPD) patients meeting all selection criteria from the United States (US) IBM MarketScan database (contained data collected from January 1, 2008 to March 31, 2018).
- UK CPRD GOLD - Overall: All chronic obstructive pulmonary disease (COPD) patients meeting all selection criteria from the United Kingdom (UK) CPRD GOLD database (contained data collected from November 21, 1987 to June 30, 2018).
Period: Overall Study
Arm/Group | US IBM Marketscan - Overall | UK CPRD GOLD - Overall
Started | 1280486 | 90660
Completed | 1280486 | 90660
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan (contained data collected from January 1, 2008 to March 31, 2018) and the United Kingdom (UK) CPRD GOLD databases (contained data collected from November 21, 1987 to June 30, 2018).
Groups:
- Total: Total of all reporting groups
Arm/Group | US IBM Marketscan - Overall | UK CPRD GOLD - Overall | Total
Number analyzed (Participants) | 1280486 | 90660 | 1371146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (13.2) | 65.9 (13.5) | 65.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 649296 | 46923 | 696219
  Male | 631190 | 43737 | 674927
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Age of the Chronic Obstructive Pulmonary Disease (COPD) Patients at the Time of COPD Diagnosis - US
Description: Age of the chronic obstructive pulmonary disease (COPD) patients at the time of COPD diagnosis from the United States (US) IBM MarketScan was reported by groups stratified according to their COPD diagnosis times (Before versus after the approval of Tiotropium + Olodaterol in 2015).
Time Frame: At index date of cohort entry (baseline; time of COPD diagnosis).
Population: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database (contained data collected from January 1, 2008 to March 31, 2018).
Measure: Mean (Standard Deviation); unit: Years
Groups:
- US IBM Marketscan - COPD Diagnosis Before Tio+Olo Approval: Cohort of chronic obstructive pulmonary disease (COPD) patients meeting all selection criteria from the United States (US) IBM MarketScan database (contained data collected from January 1, 2008 to March 31, 2018).
  Only patients who were diagnosed COPD before the approval of Tiotropium + Olodaterol (Tio+Olo) in 21 May 2015 were included in this group.
- US IBM Marketscan - COPD Diagnosis After Tio+Olo Approval: Cohort of chronic obstructive pulmonary disease (COPD) patients meeting all selection criteria from the United States (US) IBM MarketScan database (contained data collected from January 1, 2008 to March 31, 2018).
  Only patients who were diagnosed COPD after the approval of Tiotropium + Olodaterol (Tio+Olo) in 21 May 2015 were included in this group.
Arm/Group | US IBM Marketscan - COPD Diagnosis Before Tio+Olo Approval | US IBM Marketscan - COPD Diagnosis After Tio+Olo Approval
Number analyzed (Participants) | 1021963 | 258523
Years | 65.6 (13.3) | 64.4 (12.8)

2. Primary Outcome: Age of the Chronic Obstructive Pulmonary Disease (COPD) Patients at the Time of COPD Diagnosis - UK
Description: Age of the chronic obstructive pulmonary disease (COPD) patients at the time of COPD diagnosis from the the United Kingdom (UK) CPRD GOLD database was reported by groups stratified according to their COPD diagnosis times (Before versus after the approval of Tiotropium + Olodaterol in 2015).
Time Frame: At index date of cohort entry (baseline; time of COPD diagnosis).
Population: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database (contained data collected from November 21, 1987 to June 30, 2018).
Measure: Mean (Standard Deviation); unit: Years
Groups:
- UK CPRD GOLD - COPD Diagnosis Before Tio+Olo Approval: Cohort of chronic obstructive pulmonary disease (COPD) patients meeting all selection criteria from the United Kingdom (UK) CPRD GOLD database (contained data collected from November 21, 1987 to June 30, 2018).
  Only patients who were diagnosed COPD before the approval of Tiotropium + Olodaterol (Tio+Olo) in 1 July 2015 were included in this group.
- UK CPRD GOLD - COPD Diagnosis After Tio+Olo Approval: Cohort of chronic obstructive pulmonary disease (COPD) patients meeting all selection criteria from the United Kingdom (UK) CPRD GOLD database (contained data collected from November 21, 1987 to June 30, 2018).
  Only patients who were diagnosed COPD after the approval of Tiotropium + Olodaterol (Tio+Olo) in 1 July 2015 were included in this group.
Arm/Group | UK CPRD GOLD - COPD Diagnosis Before Tio+Olo Approval | UK CPRD GOLD - COPD Diagnosis After Tio+Olo Approval
Number analyzed (Participants) | 79412 | 11248
Years | 65.82 (13.81) | 66.17 (11.17)

3. Primary Outcome: Charlson Comorbidity Index (CCI) at the Time of COPD Diagnosis
Description: The Charlson Comorbidity Index (CCI) was a method of categorizing comorbidities of patients based on the International Classification of Diseases diagnosis. The CCI score ranged from 0 (better outcome) to 21 (worse outcome). The higher the score, the more fragile/ill the patient was.
Time Frame: At index date of cohort entry (baseline; time of COPD diagnosis).
Population: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan (contained data collected from January 1, 2008 to March 31, 2018) and the United Kingdom (UK) CPRD GOLD databases (contained data collected from November 21, 1987 to June 30, 2018). Results were reported by overall and by stratified groups according to Tiotropium + Olodaterol approval date for US and UK datasets, respectively.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | US IBM Marketscan - Overall | US IBM Marketscan - COPD Diagnosis Before Tio+Olo Approval | US IBM Marketscan - COPD Diagnosis After Tio+Olo Approval | UK CPRD GOLD - Overall | UK CPRD GOLD - COPD Diagnosis Before Tio+Olo Approval | UK CPRD GOLD - COPD Diagnosis After Tio+Olo Approval
Number analyzed (Participants) | 1280486 | 1021963 | 258523 | 90660 | 79412 | 11248
Score on a scale | 1.6 (1.9) | 1.5 (1.9) | 1.9 (2.1) | 1.89 (1.38) | 1.83 (1.32) | 2.31 (1.66)

4. Primary Outcome: Age of Patients Receiving First Maintenance Treatment - US
Description: Age of chronic obstructive pulmonary disease (COPD) patients initiated their first maintenance therapy in the United States (US) IBM MarketScan database was reported.
Time Frame: At index date of the first maintenance treatment
Population: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database (contained data collected from January 1, 2008 to March 31, 2018) initiated their first maintenance therapy at the time of or after the launch date of Sp(t)iolto (referred to as Tiotropium + Olodaterol; 21 May 2015), and were free from asthma. Results were reported by overall and by stratified groups according to therapies.
Measure: Mean (Inter-Quartile Range); unit: Years
Groups:
- US IBM Marketscan - 1MT - Overall: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
- US IBM Marketscan - 1MT - ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Inhaled Corticosteroid (ICS) were included in this group.
- US IBM Marketscan - 1MT - LABA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Beta-Agonists (LABA) were included in this group.
- US IBM Marketscan - 1MT - LABA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Beta-Agonists + Inhaled Corticosteroid (LABA+ICS) were included in this group.
- US IBM Marketscan - 1MT - LAMA+LABA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Beta-Agonists + Long-Acting Muscarinic Antagonists (LABA+LAMA) were included in this group.
- US IBM Marketscan - 1MT - LAMA+LABA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Muscarinic Antagonists + Long-Acting Beta-Agonists + Inhaled Corticosteroid (LAMA+LABA+ICS) were included in this group.
- US IBM Marketscan - 1MT - LAMA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Muscarinic Antagonists (LAMA) were included in this group.
- US IBM Marketscan - 1MT - LAMA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Muscarinic Antagonists + Inhaled Corticosteroid (LAMA+ICS) were included in this group
Arm/Group | US IBM Marketscan - 1MT - Overall | US IBM Marketscan - 1MT - ICS | US IBM Marketscan - 1MT - LABA | US IBM Marketscan - 1MT - LABA+ICS | US IBM Marketscan - 1MT - LAMA+LABA | US IBM Marketscan - 1MT - LAMA+LABA+ICS | US IBM Marketscan - 1MT - LAMA | US IBM Marketscan - 1MT - LAMA+ICS
Number analyzed (Participants) | 53473 | 6737 | 351 | 26378 | 6745 | 2237 | 10892 | 133
Years | 63.0 [57.0 to 73.0] | 62.0 [56.0 to 73.0] | 67.0 [59.0 to 79.0] | 62.0 [56.0 to 72.0] | 62.0 [56.0 to 72.0] | 63.0 [58.0 to 74.0] | 64.0 [58.0 to 75.0] | 65.0 [58.0 to 76.0]

5. Primary Outcome: Charlson Comorbidity Index (CCI) of Patients Receiving First Maintenance Treatment - US
Description: as for outcome 3
Time Frame: At index date of the first maintenance treatment
Population: as for outcome 4
Measure: Mean (Inter-Quartile Range); unit: Score on a scale
Arm/Group | US IBM Marketscan - 1MT - Overall | US IBM Marketscan - 1MT - ICS | US IBM Marketscan - 1MT - LABA | US IBM Marketscan - 1MT - LABA+ICS | US IBM Marketscan - 1MT - LAMA+LABA | US IBM Marketscan - 1MT - LAMA+LABA+ICS | US IBM Marketscan - 1MT - LAMA | US IBM Marketscan - 1MT - LAMA+ICS
Number analyzed (Participants) | 53473 | 6737 | 351 | 26378 | 6745 | 2237 | 10892 | 133
Score on a scale | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0]

6. Primary Outcome: Characteristics of Patients Receiving First Maintenance Treatment - US
Description: Characteristics of patients receiving first maintenance treatment among chronic obstructive pulmonary disease (COPD) patients initiated their first maintenance therapy in the United States (US) IBM MarketScan database were reported.
Time Frame: At index date of the first maintenance treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | US IBM Marketscan - 1MT - Overall | US IBM Marketscan - 1MT - ICS | US IBM Marketscan - 1MT - LABA | US IBM Marketscan - 1MT - LABA+ICS | US IBM Marketscan - 1MT - LAMA+LABA | US IBM Marketscan - 1MT - LAMA+LABA+ICS | US IBM Marketscan - 1MT - LAMA | US IBM Marketscan - 1MT - LAMA+ICS
Number analyzed (Participants) | 53473 | 6737 | 351 | 26378 | 6745 | 2237 | 10892 | 133
Participants
  Upper respiratory tract infection | 13803 | 2114 | 87 | 7151 | 1632 | 486 | 2299 | 34
  Lower respiratory tract infection | 8525 | 1160 | 46 | 4577 | 885 | 367 | 1474 | 16
  Pneumonia | 9946 | 1253 | 77 | 4762 | 1014 | 651 | 2160 | 29
  Chronic bronchitis | 5161 | 603 | 42 | 2642 | 502 | 294 | 1066 | 12
  Lung fibrosis | 1868 | 239 | 22 | 882 | 207 | 108 | 405 | 5
  Concomitant medications - Oral corticosteroids | 23272 | 3172 | 152 | 12240 | 2770 | 929 | 3959 | 50
  Concomitant medications - Oral antibiotics | 37829 | 5047 | 249 | 19168 | 4645 | 1508 | 7116 | 96
  Concomitant medications - Oxygen therapy | 4580 | 425 | 57 | 2094 | 625 | 305 | 1058 | 16

7. Primary Outcome: Age of Patients Receiving First Maintenance Treatment - UK
Description: Age of patients receiving first maintenance treatment from chronic obstructive pulmonary disease (COPD) patients initiated their first maintenance therapy in the United Kingdom (UK) CPRD GOLD database was reported.
Time Frame: At index date of the first maintenance treatment
Population: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database (contained data collected from November 21, 1987 to June 30, 2018) initiated their first maintenance therapy at the time of or after the launch date of Sp(t)iolto (referred to as Tiotropium+Olodaterol; 1 July 2015), and were free from asthma. Results were reported by overall and by stratified groups according to therapies.
Measure: Median (Inter-Quartile Range); unit: Years
Groups:
- UK CPRD GOLD - 1MT - Overall: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
- UK CPRD GOLD - 1MT - ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Inhaled Corticosteroid (ICS) were included in this group.
- UK CPRD GOLD - 1MT - LABA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Beta-Agonists (LABA) were included in this group.
- UK CPRD GOLD - 1MT - LABA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Beta-Agonists + Inhaled Corticosteroid (LABA+ICS) were included in this group.
- UK CPRD GOLD - 1MT - LAMA+LABA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Beta-Agonists + Long-Acting Muscarinic Antagonists (LABA+LAMA) were included in this group.
- UK CPRD GOLD - 1MT - LAMA+LABA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Muscarinic Antagonists + Long-Acting Beta-Agonists + Inhaled Corticosteroid (LAMA+LABA+ICS) were included in this group.
- UK CPRD GOLD - 1MT - LAMA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Muscarinic Antagonists (LAMA) were included in this group.
- UK CPRD GOLD - 1MT - LAMA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Muscarinic Antagonists + Inhaled Corticosteroid (LAMA+ICS) were included in this group.
Arm/Group | UK CPRD GOLD - 1MT - Overall | UK CPRD GOLD - 1MT - ICS | UK CPRD GOLD - 1MT - LABA | UK CPRD GOLD - 1MT - LABA+ICS | UK CPRD GOLD - 1MT - LAMA+LABA | UK CPRD GOLD - 1MT - LAMA+LABA+ICS | UK CPRD GOLD - 1MT - LAMA | UK CPRD GOLD - 1MT - LAMA+ICS
Number analyzed (Participants) | 8786 | 753 | 382 | 1202 | 1407 | 352 | 4675 | 15
Years | 68.0 [60.0 to 75.0] | 67.0 [59.0 to 75.0] | 67.0 [59.0 to 75.0] | 67.0 [59.0 to 75.0] | 68.0 [61.0 to 75.0] | 70.0 [62.0 to 77.0] | 68.0 [60.0 to 75.0] | 69.0 [64.0 to 73.0]

8. Primary Outcome: Characteristics of Patients Receiving First Maintenance Treatment - UK
Description: Characteristics of patients receiving first maintenance treatment from chronic obstructive pulmonary disease (COPD) patients initiated their first maintenance therapy in the United Kingdom (UK) CPRD GOLD database were reported.
Time Frame: At index date of the first maintenance treatment
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | UK CPRD GOLD - 1MT - Overall | UK CPRD GOLD - 1MT - ICS | UK CPRD GOLD - 1MT - LABA | UK CPRD GOLD - 1MT - LABA+ICS | UK CPRD GOLD - 1MT - LAMA+LABA | UK CPRD GOLD - 1MT - LAMA+LABA+ICS | UK CPRD GOLD - 1MT - LAMA | UK CPRD GOLD - 1MT - LAMA+ICS
Number analyzed (Participants) | 8786 | 753 | 382 | 1202 | 1407 | 352 | 4675 | 15
Participants
  Upper respiratory tract infection | 3802 | 454 | 166 | 545 | 541 | 143 | 1946 | 7
  Lower respiratory tract infection (not pneumonia) | 4835 | 501 | 220 | 721 | 732 | 164 | 2486 | 11
  Concomitant medications - Oral corticosteroids | 2367 | 207 | 87 | 453 | 353 | 121 | 1140 | 6
  Concomitant medications - Oral antibiotics | 5133 | 480 | 204 | 796 | 797 | 224 | 2624 | 8

9. Primary Outcome: Age of Patients Receiving Second Maintenance Treatment - US
Description: Age of patients receiving second maintenance treatment from the United States (US) IBM MarketScan database was reported.
Time Frame: At index date of the second maintenance treatment
Population: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database (contained data collected from January 1, 2008 to March 31, 2018) initiated their second maintenance therapy and were free from asthma prior to initiation of first maintenance therapy. Results were reported by overall and by stratified groups according to therapies.
Measure: Median (Inter-Quartile Range); unit: Years
Groups:
- US IBM Marketscan - 2MT - Overall: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy (2MT) and were free from asthma prior to initiation of first maintenance therapy.
- US IBM Marketscan - 2MT - ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy (2MT) and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Inhaled Corticosteroid (ICS) were included in this group.
- US IBM Marketscan - 2MT - LABA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy (2MT) and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Long-Acting Beta-Agonists (LABA) were included in this group.
- US IBM Marketscan - 2MT - LABA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy (2MT) and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Long-Acting Beta-Agonists + Inhaled Corticosteroid (LABA+ICS) were included in this group.
- US IBM Marketscan - 2MT - LAMA+LABA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy (2MT) and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Long-Acting Muscarinic Antagonists + Long-Acting Beta-Agonists(LAMA+LABA) were included in this group.
- US IBM Marketscan - 2MT - LAMA+LABA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy (2MT) and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Long-Acting Muscarinic Antagonists + Long-Acting Beta-Agonists + Inhaled Corticosteroid (LAMA+LABA+ICS) were included in this group.
- US IBM Marketscan - 2MT - LAMA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy (2MT) and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Long-Acting Muscarinic Antagonists (LAMA) were included in this group.
- US IBM Marketscan - 2MT - LAMA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy (2MT) and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Long-Acting Muscarinic Antagonists + Inhaled Corticosteroid (LAMA+ICS) were included in this group.
Arm/Group | US IBM Marketscan - 2MT - Overall | US IBM Marketscan - 2MT - ICS | US IBM Marketscan - 2MT - LABA | US IBM Marketscan - 2MT - LABA+ICS | US IBM Marketscan - 2MT - LAMA+LABA | US IBM Marketscan - 2MT - LAMA+LABA+ICS | US IBM Marketscan - 2MT - LAMA | US IBM Marketscan - 2MT - LAMA+ICS
Number analyzed (Participants) | 7028 | 584 | 82 | 1813 | 1125 | 1834 | 1450 | 140
Years | 64.0 [58.0 to 74.0] | 63.0 [57.0 to 74.0] | 70.0 [62.0 to 79.0] | 63.0 [58.0 to 73.0] | 63.0 [58.0 to 73.0] | 64.0 [58.0 to 73.0] | 64.0 [59.0 to 75.0] | 65.0 [60.0 to 78.5]

10. Primary Outcome: Charlson Comorbidity Index (CCI) of Patients Receiving Second Maintenance Treatment - US
Description: as for outcome 3
Time Frame: At index date of the second maintenance treatment
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | US IBM Marketscan - 2MT - Overall | US IBM Marketscan - 2MT - ICS | US IBM Marketscan - 2MT - LABA | US IBM Marketscan - 2MT - LABA+ICS | US IBM Marketscan - 2MT - LAMA+LABA | US IBM Marketscan - 2MT - LAMA+LABA+ICS | US IBM Marketscan - 2MT - LAMA | US IBM Marketscan - 2MT - LAMA+ICS
Number analyzed (Participants) | 7028 | 584 | 82 | 1813 | 1125 | 1834 | 1450 | 140
Score on a scale | 2.0 [1.0 to 4.0] | 2.0 [2.0 to 4.0] | 3.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 5.0]

11. Primary Outcome: Characteristics of Patients Receiving Second Maintenance Treatment - US
Description: Characteristics of patients receiving second maintenance treatment from chronic obstructive pulmonary disease (COPD) patients initiated their second maintenance therapy in the United States (US) IBM MarketScan database were reported.
Time Frame: At index date of the second maintenance treatment
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | US IBM Marketscan - 2MT - Overall | US IBM Marketscan - 2MT - ICS | US IBM Marketscan - 2MT - LABA | US IBM Marketscan - 2MT - LABA+ICS | US IBM Marketscan - 2MT - LAMA+LABA | US IBM Marketscan - 2MT - LAMA+LABA+ICS | US IBM Marketscan - 2MT - LAMA | US IBM Marketscan - 2MT - LAMA+ICS
Number analyzed (Participants) | 7028 | 584 | 82 | 1813 | 1125 | 1834 | 1450 | 140
Participants
  Male | 3674 | 265 | 41 | 920 | 628 | 998 | 749 | 73
  Upper respiratory tract infection | 1842 | 196 | 25 | 497 | 307 | 442 | 343 | 32
  Lower respiratory infections | 1385 | 130 | 13 | 368 | 213 | 372 | 260 | 29
  Chronic bronchitis | 1095 | 89 | 11 | 264 | 165 | 297 | 243 | 26
  Lung fibrosis | 388 | 37 | 11 | 101 | 43 | 105 | 79 | 12
  Concomitant medications - Oral corticosteroids | 4065 | 355 | 44 | 1019 | 595 | 1125 | 851 | 75
  Concomitant medications - Oral antibiotics | 5399 | 481 | 64 | 1399 | 833 | 1388 | 1126 | 108

12. Primary Outcome: Age of Patients Receiving Second Maintenance Treatment - UK
Description: Age of patients receiving second maintenance treatment from chronic obstructive pulmonary disease (COPD) patients initiated their second maintenance therapy in the United Kingdom (UK) CPRD GOLD database was reported.
Time Frame: At index date of the second maintenance treatment
Population: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database (contained data collected from November 21, 1987 to June 30, 2018) initiated their second maintenance therapy at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma prior to initiation of first maintenance therapy. Results were reported by overall and by stratified groups according to therapies.
Measure: Median (Inter-Quartile Range); unit: Years
Groups:
- UK CPRD GOLD - 2MT - Overall: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their second maintenance therapy (2MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma prior to initiation of first maintenance therapy.
- UK CPRD GOLD - 2MT - ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their second maintenance therapy (2MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Inhaled Corticosteroid (ICS) were included in this group.
- UK CPRD GOLD - 2MT - LABA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their second maintenance therapy (2MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Beta-Agonists (LABA) were included in this group.
- UK CPRD GOLD - 2MT - LABA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their second maintenance therapy (2MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Beta-Agonists + Inhaled Corticosteroid (LABA+ICS) were included in this group.
- UK CPRD GOLD - 2MT - LAMA+LABA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their second maintenance therapy (2MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Beta-Agonists + Long-Acting Muscarinic Antagonists (LABA+LAMA) were included in this group.
- UK CPRD GOLD - 2MT - LAMA+LABA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their second maintenance therapy (2MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Muscarinic Antagonists + Long-Acting Beta-Agonists + Inhaled Corticosteroid (LAMA+LABA+ICS) were included in this group.
- UK CPRD GOLD - 2MT - LAMA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their second maintenance therapy (2MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Muscarinic Antagonists (LAMA) were included in this group.
- UK CPRD GOLD - 2MT - LAMA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United Kingdom (UK) CPRD GOLD database initiated their first maintenance therapy (1MT) at the time of or after the launch date of Tiotropium + Olodaterol, and were free from asthma.
  Only patients who were treated with Long-Acting Muscarinic Antagonists + Inhaled Corticosteroid (LAMA+ICS) were included in this group.
Arm/Group | UK CPRD GOLD - 2MT - Overall | UK CPRD GOLD - 2MT - ICS | UK CPRD GOLD - 2MT - LABA | UK CPRD GOLD - 2MT - LABA+ICS | UK CPRD GOLD - 2MT - LAMA+LABA | UK CPRD GOLD - 2MT - LAMA+LABA+ICS | UK CPRD GOLD - 2MT - LAMA | UK CPRD GOLD - 2MT - LAMA+ICS
Number analyzed (Participants) | 2461 | 60 | 101 | 338 | 970 | 685 | 222 | 85
Years | 68.0 [61.0 to 75.0] | 68.0 [61.5 to 74.0] | 71.0 [63.0 to 76.0] | 69.0 [61.0 to 77.0] | 68.0 [61.0 to 74.0] | 68.0 [60.0 to 74.0] | 70.0 [62.0 to 77.0] | 68.0 [59.0 to 73.0]

13. Primary Outcome: Characteristics of Patients Receiving Second Maintenance Treatment - UK
Description: Characteristics of patients receiving second maintenance treatment from chronic obstructive pulmonary disease (COPD) patients initiated their second maintenance therapy in the United Kingdom (UK) CPRD GOLD database were reported.
Time Frame: At index date of the second maintenance treatment
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | UK CPRD GOLD - 2MT - Overall | UK CPRD GOLD - 2MT - ICS | UK CPRD GOLD - 2MT - LABA | UK CPRD GOLD - 2MT - LABA+ICS | UK CPRD GOLD - 2MT - LAMA+LABA | UK CPRD GOLD - 2MT - LAMA+LABA+ICS | UK CPRD GOLD - 2MT - LAMA | UK CPRD GOLD - 2MT - LAMA+ICS
Number analyzed (Participants) | 2461 | 60 | 101 | 338 | 970 | 685 | 222 | 85
Participants
  Male | 1375 | 31 | 51 | 191 | 555 | 383 | 127 | 37
  Concomitant medications - Oral corticosteroids | 1066 | 25 | 36 | 152 | 356 | 385 | 71 | 41

14. Secondary Outcome: Number of Participants With Zero Exacerbations in the Year Prior to the Start of First Maintenance Therapy - US
Description: Number of participants with zero exacerbations in the year prior to the start of first maintenance therapy among the chronic obstructive pulmonary disease (COPD) patients initiated their first maintenance therapy the United States (US) IBM MarketScan database was reported.
Time Frame: At index date of the first maintenance treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | US IBM Marketscan - 1MT - Overall | US IBM Marketscan - 1MT - ICS | US IBM Marketscan - 1MT - LABA | US IBM Marketscan - 1MT - LABA+ICS | US IBM Marketscan - 1MT - LAMA+LABA | US IBM Marketscan - 1MT - LAMA+LABA+ICS | US IBM Marketscan - 1MT - LAMA | US IBM Marketscan - 1MT - LAMA+ICS
Number analyzed (Participants) | 53473 | 6737 | 351 | 26378 | 6745 | 2237 | 10892 | 133
Participants | 26242 | 3518 | 183 | 12483 | 3818 | 676 | 5515 | 49

15. Secondary Outcome: Number of Participants With Zero Exacerbations in the Year Prior to the Start of First Maintenance Therapy - UK
Description: Number of participants with zero exacerbations in the year prior to the start of first maintenance therapy among the chronic obstructive pulmonary disease (COPD) patients initiated their first maintenance therapy in the United Kingdom (UK) CPRD GOLD database was reported.
Time Frame: At index date of the first maintenance treatment
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | UK CPRD GOLD - 1MT - Overall | UK CPRD GOLD - 1MT - ICS | UK CPRD GOLD - 1MT - LABA | UK CPRD GOLD - 1MT - LABA+ICS | UK CPRD GOLD - 1MT - LAMA+LABA | UK CPRD GOLD - 1MT - LAMA+LABA+ICS | UK CPRD GOLD - 1MT - LAMA | UK CPRD GOLD - 1MT - LAMA+ICS
Number analyzed (Participants) | 8786 | 753 | 382 | 1202 | 1407 | 352 | 4675 | 15
Participants | 5942 | 498 | 275 | 712 | 960 | 207 | 3281 | 9

16. Secondary Outcome: Number of Participants With Zero Exacerbations in the Year Prior to the Start of Second Maintenance Therapy - US
Description: Number of participants with zero exacerbations in the year prior to the start of second maintenance therapy among the chronic obstructive pulmonary disease (COPD) patients initiated their second maintenance therapy the United States (US) IBM MarketScan database was reported.
Time Frame: At index date of the second maintenance treatment
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Groups:
- US IBM Marketscan - 2MT - ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Inhaled Corticosteroid (ICS) were included in this group.
- US IBM Marketscan - 2MT - LABA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Long-Acting Beta-Agonists (LABA) were included in this group.
- US IBM Marketscan - 2MT - LABA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Long-Acting Beta-Agonists + Inhaled Corticosteroid (LABA+ICS) were included in this group.
- US IBM Marketscan - 2MT - LAMA+LABA+ICS: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Long-Acting Muscarinic Antagonists + Long-Acting Beta-Agonists + Inhaled Corticosteroid (LAMA+LABA+ICS) were included in this group.
- US IBM Marketscan - 2MT - LAMA: All chronic obstructive pulmonary disease (COPD) patients who meet all selection criteria from the United States (US) IBM MarketScan database initiated their second maintenance therapy and were free from asthma prior to initiation of first maintenance therapy.
  Only patients who were treated with Long-Acting Muscarinic Antagonists (LAMA) were included in this group.
Arm/Group | US IBM Marketscan - 2MT - Overall | US IBM Marketscan - 2MT - ICS | US IBM Marketscan - 2MT - LABA | US IBM Marketscan - 2MT - LABA+ICS | US IBM Marketscan - 2MT - LAMA+LABA | US IBM Marketscan - 2MT - LAMA+LABA+ICS | US IBM Marketscan - 2MT - LAMA | US IBM Marketscan - 2MT - LAMA+ICS
Number analyzed (Participants) | 7028 | 584 | 82 | 1813 | 1125 | 1834 | 1450 | 140
Participants | 2361 | 226 | 29 | 684 | 426 | 505 | 451 | 40

17. Secondary Outcome: Number of Participants With Zero Exacerbations in the Year Prior to the Start of Second Maintenance Therapy - UK
Description: Number of participants with zero exacerbations in the year prior to the start of second maintenance therapy among chronic obstructive pulmonary disease (COPD) patients initiated their second maintenance therapy in the United Kingdom (UK) CPRD GOLD database was reported.
Time Frame: At index date of the second maintenance treatment
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | UK CPRD GOLD - 2MT - Overall | UK CPRD GOLD - 2MT - ICS | UK CPRD GOLD - 2MT - LABA | UK CPRD GOLD - 2MT - LABA+ICS | UK CPRD GOLD - 2MT - LAMA+LABA | UK CPRD GOLD - 2MT - LAMA+LABA+ICS | UK CPRD GOLD - 2MT - LAMA | UK CPRD GOLD - 2MT - LAMA+ICS
Number analyzed (Participants) | 2461 | 60 | 101 | 338 | 970 | 685 | 222 | 85
Participants | 1351 | 34 | 63 | 172 | 590 | 299 | 144 | 49

18. Secondary Outcome: Days Between Index and Initiation of First Maintenance Therapy - US
Description: Days between index and initiation of first maintenance therapy among the chronic obstructive pulmonary disease (COPD) patients initiated their first maintenance therapy the United States (US) IBM MarketScan database was reported.
Time Frame: From index date until initiation of first maintenance, up to 3368 days before this study started.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | US IBM Marketscan - 1MT - Overall | US IBM Marketscan - 1MT - ICS | US IBM Marketscan - 1MT - LABA | US IBM Marketscan - 1MT - LABA+ICS | US IBM Marketscan - 1MT - LAMA+LABA | US IBM Marketscan - 1MT - LAMA+LABA+ICS | US IBM Marketscan - 1MT - LAMA | US IBM Marketscan - 1MT - LAMA+ICS
Number analyzed (Participants) | 53473 | 6737 | 351 | 26378 | 6745 | 2237 | 10892 | 133
Days | 158.0 [12.0 to 839.0] | 242.0 [17.0 to 972.0] | 233.0 [14.0 to 902.0] | 165.0 [12.0 to 833.0] | 116.0 [15.0 to 672.0] | 78.0 [7.0 to 770.0] | 136.0 [9.0 to 879.0] | 85.0 [6.0 to 957.0]

19. Secondary Outcome: Days Between Index and Initiation of First Maintenance Therapy - UK
Description: Days between index and initiation of first maintenance therapy among the chronic obstructive pulmonary disease (COPD) patients initiated their first maintenance therapy in the United Kingdom (UK) CPRD GOLD database were reported.
Time Frame: From index date until initiation of first maintenance therapy, up to 9795 days before this study started.
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | UK CPRD GOLD - 1MT - Overall | UK CPRD GOLD - 1MT - ICS | UK CPRD GOLD - 1MT - LABA | UK CPRD GOLD - 1MT - LABA+ICS | UK CPRD GOLD - 1MT - LAMA+LABA | UK CPRD GOLD - 1MT - LAMA+LABA+ICS | UK CPRD GOLD - 1MT - LAMA | UK CPRD GOLD - 1MT - LAMA+ICS
Number analyzed (Participants) | 8786 | 753 | 382 | 1202 | 1407 | 352 | 4675 | 15
Days | 28.5 [1.0 to 521.0] | 708.0 [43.0 to 3145.0] | 43.5 [1.0 to 555.0] | 32.0 [1.0 to 566.0] | 19.0 [1.0 to 368.0] | 19.0 [1.0 to 141.5] | 22.0 [1.0 to 376.0] | 19.0 [1.0 to 123.0]

20. Secondary Outcome: Days Between First and Second Maintenance Therapy - US
Description: Days between first and second maintenance therapy among the chronic obstructive pulmonary disease (COPD) patients initiated their second maintenance therapy the United States (US) IBM MarketScan database were reported.
Time Frame: From the index date of first maintenance initiation until the initiation of the second maintenance therapy, up to 1020 days before this study started.
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | US IBM Marketscan - 2MT - Overall | US IBM Marketscan - 2MT - ICS | US IBM Marketscan - 2MT - LABA | US IBM Marketscan - 2MT - LABA+ICS | US IBM Marketscan - 2MT - LAMA+LABA | US IBM Marketscan - 2MT - LAMA+LABA+ICS | US IBM Marketscan - 2MT - LAMA | US IBM Marketscan - 2MT - LAMA+ICS
Number analyzed (Participants) | 7028 | 584 | 82 | 1813 | 1125 | 1834 | 1450 | 140
Days | 160.0 [76.0 to 335.0] | 181.5 [89.5 to 339.5] | 176.0 [86.0 to 282.0] | 158.0 [74.0 to 321.0] | 223.0 [100.0 to 415.0] | 143.5 [70.0 to 314.0] | 137.0 [66.0 to 301.0] | 125.0 [67.0 to 266.5]

21. Secondary Outcome: Days Between First and Second Maintenance Therapy - UK
Description: Days between first and second maintenance therapy among chronic obstructive pulmonary disease (COPD) patients initiated their second maintenance therapy in the United Kingdom (UK) CPRD GOLD database were reported.
Time Frame: From the index date of first maintenance initiation until the initiation of the second maintenance therapy, up to 10133 days before this study started.
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | UK CPRD GOLD - 2MT - Overall | UK CPRD GOLD - 2MT - ICS | UK CPRD GOLD - 2MT - LABA | UK CPRD GOLD - 2MT - LABA+ICS | UK CPRD GOLD - 2MT - LAMA+LABA | UK CPRD GOLD - 2MT - LAMA+LABA+ICS | UK CPRD GOLD - 2MT - LAMA | UK CPRD GOLD - 2MT - LAMA+ICS
Number analyzed (Participants) | 2461 | 60 | 101 | 338 | 970 | 685 | 222 | 85
Days | 218.0 [86.0 to 428.0] | 239.5 [61.5 to 528.0] | 141.0 [74.0 to 412.0] | 155.5 [67.0 to 335.0] | 284.0 [113.0 to 483.0] | 197.0 [82.0 to 397.0] | 225.5 [96.0 to 415.0] | 158.0 [71.0 to 281.0]

ADVERSE EVENTS:
Description: This study was based on the use of secondary data without access to individual patient data. Adverse events were not collected. Zeros in the numbers of participants at risk and affected in the "All-Cause Mortality", "Serious Adverse Events", and "Other Adverse Events" sections stand for adverse event was not collected and not available for this study.
Arm/Group | US IBM Marketscan - Overall | UK CPRD GOLD - Overall
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT04926233/Prot_SAP_000.pdf